CLINICAL TRIAL: NCT04935541
Title: The Comparison of Dexmedetomidine and Remifentanil Infusion in Geriatric Patients Undergoing Outpatient Cataract Surgery: A Prospective, Randomized, Blinded Study
Brief Title: Dexmedetomidine vs. Remifentanil Undergoing Cataract Surgery in Geriatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HEK 09/59-19
Record Dates: First submitted 2021-06-07; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Geriatrics; Outpatients; Personal Satisfaction
Keywords: geriatrics; ambulatory surgery; cataract; anesthesia; conscious sedation; dexmedetomidine; remifentanil
MeSH Terms: conditions — Personal Satisfaction; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The surgeon who performed the surgery, the participants included in the study, and the technician who collected the study data were unaware of the study groups and the type of drugs used for sedation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine infusion (Active Comparator): Dexmedetomidine (Precedex, Meditera, USA) was administered at a loading dose of 1 µg/kg for 10 minutes before local anesthesia to be applied to the eye by the surgeon. During the surgical procedure, it was administered at a dose of 0.4 µg/kg/h-1 infusion.
  Interventions: Drug: Dexmedetomidine infusion
- Remifentanil infusion (Active Comparator): Remifentanil (Ultiva, Glaxo SmithKline, Turkey) infusion was started at a dose of 0.05 µg/kg/min-1, 10 minutes before the start of the surgery as baseline infusion and continued at the same infusion dose throughout the surgical procedure.
  Interventions: Drug: Remifentanil infusion

INTERVENTIONS:
Drug: Dexmedetomidine infusion — After Dexmedetomidine infusion was given for 10 minutes, local anesthesia was applied by the surgeon. Peribulbar block and periorbital infiltration application were performed by applying a mixture of lidocaine (Jetokain, Adeka, Turkey) and 1/200000 adrenaline. After the local anesthetic agent was applied by the surgeon, orbital compression was provided for 5 minutes with maximum pressure to block the eyelid movements. Cataract surgery procedures of all patients included in the study were performed by the same surgeon.
  Other Names: Cataract surgery
  Arms: Dexmedetomidine infusion
Drug: Remifentanil infusion — After Remifentanil infusion was given for 10 minutes, local anesthesia was applied by the surgeon. Peribulbar block and periorbital infiltration application were performed by applying a mixture of lidocaine (Jetokain, Adeka, Turkey) and 1/200000 adrenaline. After the local anesthetic agent was applied by the surgeon, orbital compression was provided for 5 minutes with maximum pressure to block the eyelid movements. Cataract surgery procedures of all patients included in the study were performed by the same surgeon.
  Other Names: Cataract surgery
  Arms: Remifentanil infusion

SUMMARY:
Dexmedetomidine is an α2-adrenergic receptor agonist used for its sympatholytic effect, providing sedation, analgesia, and cardiovascular stabilization in the perioperative period. Remifentanil is a µ opioid agonist with a rapid onset and short duration of action, which is degraded by plasma esterase in tissues. Investigators aimed to compare the effects of dexmedetomidine and remifentanil infusions on sedation quality, side effects, and surgeon's satisfaction in geriatric outpatients who underwent cataract surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is an α2 agonist and remifentanil is a short-acting μ, opioid agonist. The aim of this study was to compare dexmedetomidine and remifentanil infusions used for conscious sedation in geriatric patients undergoing outpatient cataract surgery in terms of sedation quality, hemodynamic stability, and surgeon satisfaction.

Eighty patients were divided into two groups according to the administration of dexmedetomidine (Group D) and remifentanil (Group R) infusion in this randomized, prospective, double-blinded study. In group D (n = 40), after a loading of 1 µg/kg dexmedetomidine in 10 minutes, 0.4 µg/kg/h-1 infusion was administered. In Group R (n = 40), remifentanil at a dose of 0.05 µg/kg-1 was administered for 10 minutes, and then 0.05 µg/kg/min-1 infusion was continued.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 65-80,
* Who will undergo cataract surgery,
* With the American Society of Anesthesiologists (ASA) score I-III.

Exclusion Criteria:

* Second or third-degree heart block,
* Chronic α2-agonist use,
* Inability to communicate with the patient,
* Uncontrolled systemic disease,
* Allergy to local anesthetics,
* Chronic analgesic or sedative drug use,
* History of alcohol or substance addiction.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Patients between the ages of 65-80 were enrolled in the study.
Enrollment: 80 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sedation quality | Time interval immediately after the start of the surgery and before the patient is transferred to the postoperative care unit.
  The Observer Assessment Warning/Sedation Scale (OAA/S) was used to determine the sedation quality of each patient. The minimum and maximum values of OAA/S scale was between 0 and 5. Lower scores mean a better sedation quality.
Sedation level | The time interval immediately after the surgery starts and immediately after the surgery ends.
  Bispectral Index (BIS) was used to determine the sedation level of each patient. The minimum and maximum values for BIS were between 0 and 100. Lower scores mean a deep sedation level.
Pain intensity | The time interval between the start of the surgery and the end of the surgery.
  The Verbal Rating Scale was used to determine severity of the pain in the perioperative period. VRS is a 5-point scale including expressions defining the level of pain intensity (no pain, mild pain, moderate pain, intense pain and maximum pain). Higher scores mean intense pain.

SECONDARY OUTCOMES:
Side effects | The time interval between the start and the end of the surgery.
  The Vissual Analogue Scale (VAS) was used to measure the frequency and severity of nausea and vomiting in the perioperative period. The VAS score is discovered by measuring the distance (mm) on the 100-mm line. Patients scoring 75 mm or more were considered to have clinically significant nausea and vomiting.
Surgeon's satisfaction | Immediately after the surgeon finishes the operation.
  The surgeon's satisfaction in terms of the patient's sedation level, cooperation, and anesthesia management was evaluated using a questionnaire. The clinician satisfaction questionnaire was also classified as follows; 0: Not satisfied, 1: Less Satisfied, 2: Satisfied.
Pain intensity | Immediately after the surgical procedure is completed and the patient is transferred to the postoperative care unit and before the patient is transferred to the outpatient service.
  The Visual Analogue Scale (VAS) was used to determine the pain intensity in the postoperative period. The pain score is discovered by measuring the distance (mm) on the 100-mm line. Pain level was classified as follows; no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Nalan Celebi, Professor, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We plan to share our patients' data and statistical analysis with individual researchers.

REFERENCES:
- [Background] Kumar CM, Seet E, Eke T, Irwin MG, Joshi GP. Peri-operative considerations for sedation-analgesia during cataract surgery: a narrative review. Anaesthesia. 2019 Dec;74(12):1601-1610. doi: 10.1111/anae.14845. Epub 2019 Sep 19. PMID 31535721